CLINICAL TRIAL: NCT01438515
Title: Randomized Controlled Trial of Chlorhexidine Gluconate, Intranasal Mupirocin, Rifampin and Doxycycline Versus Chlorhexidine Gluconate and Intranasal Mupirocin Alone for the Eradication of Methicillin-resistant Staphylococcus Aureus Among an Ambulatory Patient Population
Brief Title: Randomized Controlled Trial of Standard Versus Systemic Decolonization Therapy for the Eradication of Methicillin-resistant Staphylococcus Aureus (MRSA) Colonization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Duncan Webster, Physician, Infectious Diseases and Medical Microbiology, Horizon Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-1265
Record Dates: First submitted 2011-09-21; First posted 2011-09-22 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Methicillin-resistant Staphylococcus Aureus
Keywords: MRSA; doxycycline; rifampin; mupirocin; chlorhexidine gluconate; decolonization; methicillin-resistant staphylococcus aureus
MeSH Terms: interventions — Rifampin; Doxycycline; chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systemic decolonization (Experimental): 7-day course of 4% chlorhexidine gluconate daily washes and 2% mupirocin ointment to the anterior nares twice daily in addition to oral rifampin (600mg daily), and doxycycline (100mg twice daily)
  Interventions: Drug: Rifampin; Drug: Doxycycline; Other: 2% mupirocin ointment; Other: 4% chlorhexidine gluconate
- Standard decolonization (Active Comparator): 7-day course of 2% mupirocin ointment to the anterior nares twice daily and 4% chlorhexidine gluconate washes once per day.
  Interventions: Other: 2% mupirocin ointment; Other: 4% chlorhexidine gluconate

INTERVENTIONS:
Drug: Rifampin — 600mg po once daily x 7 days
  Arms: Systemic decolonization
Drug: Doxycycline — 100mg po twice daily x 7 days
  Arms: Systemic decolonization
Other: 2% mupirocin ointment — ~ 1cm applied to the anterior nares twice daily for 7 days
Other: 4% chlorhexidine gluconate — Daily full body wash (including hair) for 7 days

SUMMARY:
MRSA decolonization may reduce the risk of subsequent MRSA infection and further transmission. A recent randomized controlled trial demonstrated that systemic decolonization may be safe and effective among hospitalized patients when compared to no treatment. As a large number of the investigators patients require re-admission and further transmission may take place in the community, the investigators are comparing the standard decolonization protocol for MRSA eradication to the systemic decolonization protocol among an ambulatory population.

Standard decolonization protocols, which use only topical agents, are limited in efficacy. The method of systemic decolonization to be studied here appears to have greater efficacy than the standard approach using only topical agents. However, concerns have been raised that the increased use of systemic antibiotics may lead to increased levels of drug resistance adverse effects, without sustained decolonization. This study seeks to provide further data to help answer these questions and provide guidance for further policy development and implementation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient colonized with MRSA

Exclusion Criteria:

* Currently on treatment with antibiotics
* Pregnant or breastfeeding women
* Active infection
* Hepatic cirrhosis or abnormal INR due to liver disease
* Decolonization in the previous two (2) months
* MRSA bacteria resistant to one or more of the study medications
* AST and ALT levels more than five times the upper limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of sustained decolonization at 1 month, 3 months, 6 months and 12 months | 12 months
  To compare standard versus systemic decolonization for their ability to sustain MRSA decolonization up to one year post-decolonization.

SECONDARY OUTCOMES:
Changes in susceptibility patterns of MRSA isolates. | 12 months
  Study isolates will be evaluated with regards to mupirocin, rifampin and tetracycline resistance patterns, where individuals remain colonized, or re-colonize subsequent to implementation of the decolonization protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Webster, MA, MD, Principal Investigator — Horizon Health Network
Locations (1):
- Saint John Regional Hospital, Saint John, New Brunswick, Canada

REFERENCES:
- [Background] Simor AE, Phillips E, McGeer A, Konvalinka A, Loeb M, Devlin HR, Kiss A. Randomized controlled trial of chlorhexidine gluconate for washing, intranasal mupirocin, and rifampin and doxycycline versus no treatment for the eradication of methicillin-resistant Staphylococcus aureus colonization. Clin Infect Dis. 2007 Jan 15;44(2):178-85. doi: 10.1086/510392. Epub 2006 Dec 14. PMID 17173213